CLINICAL TRIAL: NCT03346915
Title: Integrating a Health Information Technology System With a Web-based Mobile Health Educational Intervention to Support More Effective Provider-patient Communication and HPV Vaccine Utilization
Brief Title: Integrating a Health Information Technology System for Primary and Secondary Cervical Cancer Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-36669
Record Dates: First submitted 2017-11-14; First posted 2017-11-20 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Human Papilloma Virus; Cervical Cancer; Human Papillomavirus Infection; Oropharyngeal Cancer; Vaginal Cancer; Vulvar Cancer; Anal Cancer; Penile Cancer
Keywords: HPV vaccinaton; Cervical cancer screening; Web-based mobile health education; brief negotiated interview (BNI
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections; Oropharyngeal Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Anus Neoplasms; Penile Neoplasms

STUDY DESIGN:
Intervention Model Description: We are proposing a single arm proof of concept. We will recruit 30 parents/guardians and their age-eligible child for the single arm proof of concept.
  For this proof of concept/pilot trial, we will assess the feasibility and impact of WOW to improve provider communication about HPV vaccination and increase the initial and complete vaccination rates for both boys and girls aged 9-17 and to enhance knowledge and awareness about risks and benefits of HPV vaccine among dyads. The power of our proposed pilot for determining intervention effects is limited. However, because we are proposing a proof of concept pilot and feasibility study, in our experience and that of others, our proposed sample size generally provides sufficient data to estimate subject retention, distribution of variables and feasibility as we plan for a larger-multi-site RCT of the proposed study. We expect our intervention to demonstrate feasibility of the intervention in a clinic setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects receiving WoW and BNI (Experimental): The behavioral intervention (WoW and BNI) will supplement the subject's standard of care by incorporating interactive messaging, reminders, patient education, and enhanced provider communication.
  Interventions: Behavioral: WoW and BNI

INTERVENTIONS:
Behavioral: WoW and BNI — The Text/web based health information technology system, WoW, will provide educational resources for participants and their families to learn more about HPV vaccination and cervical cancer screening. WoW will be tailored to the participant and will be based on the participant's cancer screening and HPV vaccine health needs; It will then send custom text messages based their concerns and will remind them to schedule and attend their doctor's appointment. The brief negotiated interview will encourage and empower participants to have positive behavioral changes in regards to their health.

SUMMARY:
The project aims to increase HPV vaccination and cervical cancer screening through a web-based mobile health education program called, Wheel of Wellness (WoW) and a brief negotiated interview (BNI). The in-person BNI and WoW system will provide educational resources for participants and their families to learn more about HPV vaccination and cervical cancer screening.

DETAILED DESCRIPTION:
WoW will be tailored to the participant and will be based on the participant's cancer screening and HPV vaccine health needs; It will then send custom text messages based their concerns and will remind them to schedule and attend their doctor's appointment. The researchers will conduct a single armed proof of concept where the participants will be actively using WoW. The in-person BNI will empower participants to have positive behavioral changes in regards to their health by giving them appropriate health information as well as answering their questions and concerns about cervical cancer prevention and screening.

ELIGIBILITY:
Inclusion Criteria:

1. Parent/guardian with a child between the ages of 9 to 17 who receives primary care at one of the participating sites and their male child.
2. Parent/guardian with a male child who provides consent to have child's HPV vaccination status checked in EMR.
3. Parent/guardian with a male child who has neither initiated the HPV vaccine nor completed the series
4. Parent/guardian and male child with the ability to read and write in English.
5. Parent/guardian and male child have access to a smartphone.

Exclusion Criteria:

1. Parent/guardian's eligible child is pregnant.
2. Parent/guardian's has begun or completed the HPV series.
3. Parent/guardian, in the opinion of the clinical staff, is cognitively impaired and unable to give informed consent.

Ages: 9 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
HPV vaccine series start and completion | 6 months
  The primary outcome of interest is receipt of the first dose and completion of the three-dose or two-dose series of HPV vaccine by participants within six months of intervention by EMR review.

SECONDARY OUTCOMES:
HPV and Cervical Cancer awareness and knowledge | 6-12 months
  Change in knowledge of HPV vaccination and cervical cancer will be measured using a survey, which is under development, that includes questions about HPV and HPV vaccination. It will be administered before and again after the intervention and changes in responses will be compared.
Provider-patient communication about HPV vaccine and cervical cancer | one week after provider visit throughout the duration of the study
  Based on participants' entries onto the WoW website, a list of their concerns and questions about HPV vaccine and cervical cancer will be created and this list will be brought to a clinical visit with their providers. Following the clinical visit, participants will be asked whether providers addressed their questions and concerns about HPV vaccine and cervical cancer using a short questionnaire with a 5 point likert scale where 1=completely addressed and 5= not at all addressed. Lower scores are favorable.
Wheel of Wellness (WoW) feasibility | 6 months
  The feasibility of WoW will be assessed by using a short questionnaire that measures both how easy the WoW site is to navigate and how frequently participants used the WoW site.
Wheel of Wellness (WoW) feasibility | 12 months
  The feasibility of WoW will be assessed by using a short questionnaire that measures both how easy the WoW site is to navigate and how frequently participants used the WoW site.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Joseph, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No